CLINICAL TRIAL: NCT02874131
Title: Behavioral Activation + Cognitive Processing Therapy for Posttraumatic Stress Disorder and Comorbid Major Depressive Disorder
Brief Title: Behavioral Activation + Cognitive Processing Therapy for PTSD and Comorbid MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristen Walter, Clinical Research Psychologist, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2015.0039
Record Dates: First submitted 2016-08-02; First posted 2016-08-22 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder
Keywords: Posttraumatic Stress Disorder; Major Depressive Disorder; Behavioral Activation; Cognitive Processing Therapy; Comorbidity; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Activation + CPT (Experimental): Behavioral Activation, an evidence-based treatment for depression, is combined with Cognitive Processing Therapy (CPT), an evidence-based treatment for PTSD, to address symptoms of PTSD and comorbid MDD.
  Interventions: Behavioral: Behavioral Activation; Behavioral: Cognitive Processing Therapy
- Cognitive Processing Therapy (Active Comparator): CPT is an evidence-based treatment for PTSD that has also been shown to reduce depression symptoms.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral activation
  Other Names: BA
  Arms: Behavioral Activation + CPT
Behavioral: Cognitive Processing Therapy — Cognitive processing therapy
  Other Names: CPT

SUMMARY:
This study is a randomized controlled trial comparing an integrated treatment, Behavioral Activation + Cognitive Processing Therapy (BA + CPT), to CPT alone among active-duty service members with posttraumatic stress disorder (PTSD) and comorbid major depressive disorder (MDD). Participants will complete assessor-administered and self-report measures at pre- and post-treatment assessments, as well as a 3-month follow-up. Additionally, participants will complete self-report measures of PTSD and MDD symptoms at each therapy session.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is the psychological condition most commonly comorbid with posttraumatic stress disorder (PTSD). PTSD and MDD comorbidity is associated with greater symptom severity, lower levels of functioning, greater disability, and increased suicide potential relative to PTSD or MDD alone. Unfortunately, no psychological treatment intervention specifically addresses this comorbidity. Individuals with comorbid PTSD and MDD often receive evidence-based treatments for PTSD, such as cognitive processing therapy (CPT); although such treatments typically reduce both PTSD and depression symptoms, few studies have specifically examined these outcomes in individuals with PTSD and comorbid MDD. The primary goal of this randomized controlled trial is to evaluate whether greater improvement in depression symptoms can be achieved by augmenting CPT with behavioral activation (BA), a standard depression treatment, for active-duty service members with PTSD and comorbid MDD. Participants will be evaluated at three assessment time-points (pre-treatment, post-treatment, and three-month follow-up), as well as complete self-report measures of PTSD and MDD symptoms at each therapy session.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty service member seeking mental health treatment at Naval Medical Center San Diego (NMCSD), branch clinics, or Naval Hospital Camp Pendleton (NHCP)
* Meet current diagnostic criteria for PTSD based on the DSM-5 as a consequence of any index traumatic event (e.g., combat, military sexual trauma, child abuse, accidents, etc.)
* Meet current diagnostic criteria for MDD based on DSM-5 criteria.

Exclusion Criteria:

* Unmanaged psychosis or manic episode in the past year
* Substance use disorder warranting primary substance use treatment or detoxification
* Participation in concurrent psychotherapies directly targeting PTSD
* Participation in concurrent psychotherapies directly targeting depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Prior to beginning treatment through three months following treatment completion (approximately 10 months)
  Assessor-administered measure of depression symptoms

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for the DSM-5 (CAPS-5) | Prior to beginning treatment through three months following treatment completion (approximately 10 months)
  Assessor-administered measure of PTSD symptoms
Patient Health Questionnaire (PHQ-9) | Prior to beginning treatment through three months following treatment completion (approximately 10 months)
  Self-report measure of depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: William M. Hunt, Ph.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available only in aggregate

REFERENCES:
- [Background] Walter KH, Glassman LH, Michael Hunt W, Otis NP, Thomsen CJ. Evaluation of an integrated treatment for active duty service members with comorbid posttraumatic stress disorder and major depressive disorder: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2018 Jan;64:152-160. doi: 10.1016/j.cct.2017.10.010. Epub 2017 Nov 7. PMID 29107036
- [Result] Walter KH, Hunt WM, Otis NP, Kline AC, Miggantz EL, Thomsen CJ, Glassman LH. Comparison of behavioral activation-enhanced cognitive processing therapy and cognitive processing therapy among U.S. service members: A randomized clinical trial. Psychiatry Res. 2023 Aug;326:115330. doi: 10.1016/j.psychres.2023.115330. Epub 2023 Jul 4. PMID 37418778
- [Result] Kline AC, Otis NP, Norman SB, Hunt WM, Walter KH. Dropout in a clinical trial for comorbid PTSD and MDD among US service members: Are pretreatment characteristics predictive? Psychother Res. 2025 Apr;35(4):614-626. doi: 10.1080/10503307.2024.2325519. Epub 2024 Mar 18. PMID 38497740
- [Derived] Glassman LH, Otis NP, Kline AC, Hunt WM, Walter KH. Sex differences in treatment outcomes among U.S. service members with comorbid PTSD and MDD. BMC Psychol. 2026 Jan 31. doi: 10.1186/s40359-025-03878-4. Online ahead of print. PMID 41620779
- [Derived] Otis NP, Kline AC, Glassman LH, Michael Hunt W, Walter KH. Sudden gains in cognitive processing therapy with and without behavioral activation among service members with comorbid PTSD and MDD. Behav Res Ther. 2025 Jul;190:104753. doi: 10.1016/j.brat.2025.104753. Epub 2025 Apr 22. PMID 40288269